CLINICAL TRIAL: NCT04743583
Title: Prevalence of Intrathoracic Lymph Node Calcifications and Metastatic Involvement in Patients Undergoing Endosonography for Diagnosis and/or Mediastinal Staging of Intrathoracic Malignancy: a Cross-sectional Pilot Study
Brief Title: Prevalence and Malignant Involvement of Calcified Intrathoracic Lymph Nodes in Patients Undergoing Endosonography
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3872
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-04

CONDITIONS: Lymphadenopathy; Lung Cancer; Sarcoidosis; Tuberculosis
MeSH Terms: conditions — Lymphadenopathy; Lung Neoplasms; Sarcoidosis; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endosonography group: Patients with known or suspected lung cancer or intrathoracic malignancy with indication to endosonography for diagnosis or staging of intrathoracic lymph nodes according to currently accepted international guidelines
  Interventions: Device: Endosonography B-mode examination

INTERVENTIONS:
Device: Endosonography B-mode examination — Endobronchial ultrasound (EBUS) or Endoscopic with bronchoscope (EUS-B) B-mode examination and sampling, when indicated, of lymphadenopathy

SUMMARY:
The presence of calcifications, which is a relatively common feature in intrathoracic lymph nodes, typically contributes to confer them a heterogeneous aspect during endosonographic B-mode examination, but their prevalence and a possible association between calcifications and metastatic involvement has never been systematically evaluated. We hypothesize that, in patients undergoing mediastinal diagnosis or staging of suspected/known lung cancer/intrathoracic malignancies, the prevalence of lymph node metastases is similar in calcified and non-calcified lymph nodes.

DETAILED DESCRIPTION:
The presence of calcifications, which is a relatively common feature in intrathoracic lymph nodes, typically contributes to confer them a heterogeneous aspect during endosonographic B-mode examination, but a possible association between calcifications and metastatic involvement has never been systematically evaluated. The most likely reason why this possible association has been overlooked up to now is that the presence of calcifications in intrathoracic lymph nodes has long been thought to be the consequence of the prior involvement from granulomatous diseases (i.e., tuberculosis or sarcoidosis), and as such has been considered a sign of benignity. However, the presence of lymph node calcifications at ultrasound examination is a known predictor of lymph node metastasis in patients with some specific tumours, such as the papillary thyroid carcinoma or the squamous cell carcinoma of head or neck. Furthermore, recent radiological-pathological studies have shown that metastatic foci from lung cancer are observed in up to 19% calcified mediastinal lymph nodes identified at CT in surgical candidates. Finally, a recently published EBUS study has reported, for the first time, a very strong association between a very specific pattern of mediastinal lymph node calcification, known as "starry sky sign", and metastasis from pulmonary, colonic and breast adenocarcinoma. Interestingly, the starry sky sign is characterized by the presence of few to countless dot-like calcifications which are too small to be seen at CT and can be identified only during EBUS B-mode examination.

To the best of our knowledge, no studies have been carried out to assess the correlation between the presence and the ultrasound pattern of lymph node calcifications and lymph node metastasis from lung cancer or other intrathoracic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at the time of the procedure
* Known or suspected lung cancer or other intrathoracic malignancy based on imaging (CT and/or PET/CT)
* Endosonography (EBUS and/or EUS) indicated for intrathoracic lymph node assessment/sampling according to national and international guidelines: 1) enlarged (> 1 cm on its short axis at CT) and/or PET positive lymph node; and/or 2) conditions at risk for occult mediastinal metastases, such as: i) central primary tumor; ii) primary tumor > 3 cm; iii) PET negative primary tumor; iv) ipsilateral hilar metastasis (cN1 status).

Exclusion Criteria:

* Inability or unwillingness to consent
* Compromised upper airway (i.e., concomitant head and neck cancer with upper airway obstruction; critical central airway obstruction from any cause)
* Contraindication for temporary interruption of the use of antiplatelet (excluded aspirin) or anticoagulant drugs
* American Society of Anesthesiologists grade 4

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected lung cancer or other intrathoracic malignancy with indication to endosonography for diagnosis or staging of intrathoracic lymph nodes according to currently accepted international guidelines
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
prevalence of metastatic involvement in intrathoracic lymph nodes featuring calcifications of any type | 6 months
  The prevalence of malignancy in patients with calcified intrathoracic lymph nodes will be calculated on a per lymph node basis and will be compared with the prevalence of malignancy observed in non-calcified lymph nodes

SECONDARY OUTCOMES:
The prevalence of metastatic involvement from lung cancer linked to 5 predefined patterns of lymph node calcification at B-mode ultrasound examination carried out during endosonography | 6 months
  These are the 5 patterns of calcification: a) single macrocalcification; b) multiple macrocalcifications; c) single microcalcification or local cluster of microcalcifications involving a limited area (< 20%) of the lymph node; d) few (< 10) scattered microcalcifications not distributed in a local cluster; e) countless, punctate (< 1 mm) non shadowing foci distributed across the whole lymph node (starry sky sign).
The interobserver agreement for the identification of 5 predefined patterns of lymph node calcification at endosonographic B-mode ultrasound examination | 1 month
  At the end of the study, two experienced endosonographers from different units/centers, blinded to the clinical, radiological (CT, PET) and pathological details, will be provided a video-clip of each calcified lymph node and will be asked to classify the pattern of calcification.
The prevalence of actionable mutations in the overall cohort of calcified lymph nodes identified with endosonography | 1 month
  This prevalence will be calculated on a per patient basis and will be compared with the prevalence of actionable mutations in a group of consecutive patients with non-calcified lymph nodes submitted to endosonography in the same study period and with the same indications and inclusion/exclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Catholic University of the Sacred Hearth
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No